CLINICAL TRIAL: NCT04832841
Title: IgG Antibodies After SARS-CoV-2 mRNA Vaccine in Kidney Transplantation
Brief Title: IgG Antibodies After SARS-CoV-2 mRNA Vaccine in Kidney Transplantation (TASMANIA)
Acronym: TASMANIA
Status: Completed | Type: Observational
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Prof. Ondřej Viklický, M.D., Ph.D., Head of Department of Nephrology and Transplant Center, Institute for Clinical and Experimental Medicine
Other Study IDs: G-21-07
Record Dates: First submitted 2021-04-03; First posted 2021-04-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Kidney Transplantation
Keywords: kidney transplantation; SARS-CoV-2; humoral immunity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SARS-CoV-2 naive: Kidney transplant recipients without previous SARS-CoV-2 infection verified by absence of RT-PCR test in national database who receive SARS-CoV-2 mRNA vaccine after transplantation.
  Interventions: Diagnostic Test: anti-spike SARS-CoV-2 IgG
- SARS-Cov-2 exposed: Kidney transplant recipients with previous SARS-CoV-2 exposition verified by positivity of RT-PCR test in national database who receive SARS-CoV-2 mRNA vaccine after transplantation.
  Interventions: Diagnostic Test: anti-spike SARS-CoV-2 IgG
- Waiting list: Kidney transplant recipients who were vaccinated on waiting list (a) SARS-CoV-2 naive (b) SARS-Cov-2 exposed
  Interventions: Diagnostic Test: anti-spike SARS-CoV-2 IgG

INTERVENTIONS:
Diagnostic Test: anti-spike SARS-CoV-2 IgG — Immunochemiluminescent assay by DiaSorin S.p.A. Italy

SUMMARY:
The aim of this study is to assess humoral immune response in kidney transplant recipients after SARS-CoV-2 mRNA vaccine.

DETAILED DESCRIPTION:
TASMANIA is a single-center prospective observational study with 1000 kidney transplant recipients from Institute for Clinical and Experimental Medicine (IKEM), Prague. The primary objective of the study is to assess humoral immune response to SARS-CoV-2 mRNA vaccines in SARS-CoV-2-naive kidney transplant recipients using immunochemiluminescent assay. As comparator several cohorts will be evaluated:

1. kidney transplant recipients with previous SARS-CoV-2 exposition verified by real-time reverse transcription polymerase chain reaction (RT-PCR)
2. kidney transplant recipients vaccinated on waiting list (a) SARS-CoV-2 naive (b) SARS-CoV-2 previously exposed

The secondary objective is to determine clinical variables affecting antibody levels. SARS-CoV-2 anti S1/2 antibodies will be tested ≥ 15 days after the second dose of mRNA vaccines and in 3 months after the first blood sampling.

In subanalysis 50 kidney transplant recipients will be examined for a cell-mediated immune response after SARS-CoV-2 mRNA vaccine Enzyme Linked using Immuno Spot (ELISPOT) assay.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients
* Recipient age ≥ 18 years
* Written Informed Consent and Consent for Processing Personal Data
* Vaccination with two doses of SARS-CoV-2 mRNA vaccine either before or after kidney transplantation.

Exclusion Criteria:

* Active SARS-CoV-2 infection.
* Patients that received anti-SARS-CoV-2 monoclonal antibodies.
* Active infection after vaccination
* Monoclonal antibodies treatment ahead of antibody or cellular immunity screening

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients vaccinated with 2 doses of SARS-CoV-2 mRNA vaccine either before or after kidney transplantation.
Sampling Method: Probability Sample
Enrollment: 753 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Humoral immune response in kidney transplant recipients following anti-SARS-CoV2 mRNA vaccination. | 15 days-90 days
  anti-spike SARS-CoV-2 IgG measured ≥15 days after vaccination

SECONDARY OUTCOMES:
Humoral immune response in kidney transplant recipients following anti-SARS-CoV2 mRNA vaccination. | 3 months - 6 months
  anti-spike SARS-CoV-2 IgG measured 3 ≥ months after the first blood sampling
Cellular immune response in kidney transplant recipients following anti-SARS-CoV2 mRNA vaccination. | 15 - 90 days
  Cellular immunity measured by ELISPOT assay in subgroup of 50 patients
Graft function after vaccination | 15 days-90 days
  Estimated glomerular filtration rate (eGFR)
Clinical variables affecting antibody levels | 15 days-90 days
  Sex, previous SARS-CoV-2 infection, Age, Retransplantation, BMI, time from transplant, eGFR, diabetes mellitus, use of imunosuppression (tacrolimus, cyclosporine A, CNI-free regimen, mycophenolate mofetil, depleting therapy).
The impact of frailty syndrom on humoral response in older kidney recipients (70+ years of age) following anti-SARS-CoV-2 mRNA vaccination | 15 days-90 days
  Fried frailty score

CONTACTS AND LOCATIONS:
Overall Officials: Ondrej Viklicky, Prof., Principal Investigator — Institute for Clinical and Experimental Medicine
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Czechia

REFERENCES:
- [Derived] Schmalz M, Vankova H, Rajnochova-Bloudickova S, Hruba P, Fialova M, Gurka J, Magicova M, Striz I, Zahradka I, Viklicky O. The impact of frailty syndrome on humoral response to SARS-CoV-2 mRNA vaccines in older kidney transplant recipients. Int Urol Nephrol. 2023 Nov;55(11):2959-2965. doi: 10.1007/s11255-023-03557-6. Epub 2023 Apr 7. PMID 37027078
- [Derived] Magicova M, Zahradka I, Fialova M, Neskudla T, Gurka J, Modos I, Hojny M, Raska P, Smejkal P, Striz I, Viklicky O. Determinants of Immune Response to Anti-SARS-CoV-2 mRNA Vaccines in Kidney Transplant Recipients: A Prospective Cohort Study. Transplantation. 2022 Apr 1;106(4):842-852. doi: 10.1097/TP.0000000000004044. PMID 34999659